CLINICAL TRIAL: NCT03461627
Title: Salmeterol Xinafoate and Fluticasone Propinate Powder for Inhalation for Asthma: A Randomized, Double-blind, Double-dummy, Positive-controlled, Parallel-group Trail
Brief Title: Salmeterol Xinafoate and Fluticasone Propinate Powder for Inhalation for Asthma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMTLTKS-CS-01
Record Dates: First submitted 2017-12-28; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Asthma
Keywords: randomized; double-blind; double-dummy; positive-controlled; parallel-group
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Intervention Model Description: Drug：Salmeterol Xinafoate and Fluticasone Propinate Powder for inhalation (50ug/250ug) Drug：Seretide (50ug/250ug)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salmeterol Xinafoate and Fluticasone Propinate Powder (Experimental): Salmeterol Xinafoate and Fluticasone Propinate Powder for inhalation (50ug/250ug) 50ug/250ug 1 puff twice a day for 4 weeks
  Interventions: Drug: Salmeterol Xinafoate and Fluticasone Propinate Powder
- Seretide (Active Comparator): 50ug/250ug 1 puff twice a day for 4 weeks
  Interventions: Drug: Seretide

INTERVENTIONS:
Drug: Salmeterol Xinafoate and Fluticasone Propinate Powder — 50ug/250ug 1 puff twice a day for 4 weeks
  Arms: Salmeterol Xinafoate and Fluticasone Propinate Powder
Drug: Seretide — 50ug/250ug 1 puff twice a day for 4 weeks
  Arms: Seretide

SUMMARY:
assess the efficacy and safety of Salmeterol Xinafoate and Fluticasone Propinate Powder for inhalation (50ug/250ug) in combination with seretide to patients with Asthma.

a randomized, double-blind, double-dummy, positive-controlled, parallel-group trail.

ELIGIBILITY:
Inclusion Criteria:

* Patients with asthma diagnosed according to the Global INitiative for Asthma (GINA) criteria.

  * Inadequate asthma control on an inhaled corticosteroids alone at a dose of ≤ 800 μg/day of budesonide, ≤ 1000μg/day of Beclomethasone; ≤ 500 μg/day of fluticasone
  * Inadequate asthma control on bronchodilators
  * Inadequate asthma control on an ICS (medium and low dose)-LABA combination
  * primarily diagnosed with asthma
* Positive bronchodilation test [an increase in of FEV1﹥200 ml and the FEV1 change﹥12% from the baseline] or PEF variation﹥20%
* Age between 18-70 years
* Patients should participate in the study voluntarily and sign informed consent;
* Female patients can participate if they are surgically sterile or completed menopause or females capable of having children and agree not to attempt pregnancy while receiving study therapy; Male patients can participate if they are surgically sterile or males capable of having children and agree not to attempt pregnancy while receiving study therapy.

Exclusion Criteria:

* Allergic to salmeterol, fluticasone propionate or to ventolin.
* Have a current diagnosis of chronic obstructive pulmonary disease (COPD), pneumonia, pneumothorax, atelectasis, pulmonary fibrosis, bronchopulmonary dysplasia, chronic bronchitis or other respiratory tract disorders (not including asthma).
* Any respiratory tract infection, sinus infection or eardrum infection within 4 weeks prior to the screening .visit
* History or severe cardiovascular disease or hematopoietic system disease (congestive heart failure, clinically relevant coronary heart disease, apoplexy, clinically relevant cardiac arrhythmias, aortic aneurysm, and uncontrolled hypertension (systolic blood pressure above 160mmHg or diastolic blood pressure above 100 mmHg continuously measured more than twice.))
* Patients treated with leukotriene antagonist, such as zafirlukast, pranlukast, and montelukast.
* Expected medication to improve asthma other than ventolin
* Subjects who suffer from serious, uncontrolled diseases (including psychological disorders), in researcher's opinion, under great risks.
* Hepatic dysfunction: aspartate amino transferase (AST) and alanine amino transferase (ALT) levels of > 2.0 × ULN; renal dysfunction: serum creatinine level of > ULN )
* A history of both HBV infection and HCV infection.
* In Human Immunodeficiency Virus (HIV)-positive status
* Subjects with uncontrolled diabetics or fasting glucose > 10mmol/L
* Use of any β-blocking agent, including eye-drops
* In oral glucocorticoid medication or a history of systemic corticosteroid medication within 30 days of the screening visit
* Subjects who participated in other clinical studies within 2 months
* Subjects who have previously enrolled into this study
* Pregnancy, breast-feeding or planned pregnancy during the study
* Researchers think that do not fit into the group.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline (visit 2) in Forced expiratory volume in 1 second (FEV1) on day 28 | 28 days

SECONDARY OUTCOMES:
Change from baseline (visit 2) in Forced vital capacity (FVC) on day 28 | 28 days
FEV1~AUC0-12h | 12 hours
  The Forced expiratory volume in 1 second of area under the curve from 0h to 12h on day 1
PEF | 28 days
  The mean of morning and night peak expiratory flow
The mean of morning and night Asthma symptom scores | up to 28 days
  the outcomes are respectively: Day-1~day-7,Day1~day7,Day8~day14,Day15~day21,Day22~day28
The mean of peak expiratory flow (PEF)variation of morning and night | up to 28 days
Use of ventolin during the treatment | 28 days
Number of asthma acute exacerbations with subjects | 28 days
Subject self- questionare at visit 4 | 28 days
  questionare respectively have significant effectiveness , effectiveness ,Invalid , Deterioration
Questionnaire of Asthma control test scores | 28 days
  25 score reprent Partially controlled；20-25 score represent fully controlled;<20 score represent not controlled

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong, China